CLINICAL TRIAL: NCT06692491
Title: A Phase II Clinical Study on Precision Treatment of Rare Tumours in China Guided by Patient-Derived Tumor Organoids (PDO) and Next-Generation Sequencing (NGS)
Brief Title: Study of Precision Treatment for Rare Tumours in China Guided by PDO and NGS
Acronym: SPRING
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, shubin wang, Director of Medical Oncology, Peking University Shenzhen Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUShenzhenH RE [2024]No.(117)
Record Dates: First submitted 2024-09-16; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Rare Tumour
Keywords: Rare Tumour; Patient-Derived Organoids (PDO); Next-Gneration Sequencing (NGS); Precision Treatment
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Epirubicin; Gemcitabine; Vinorelbine; Teniposide; Cisplatin; Irinotecan; Fluorouracil; Nivolumab; pembrolizumab; durvalumab; atezolizumab; sintilimab; tislelizumab; camrelizumab; toripalimab; envafolimab; osimertinib; alectinib; Vemurafenib; pamiparib; erdafitinib; pyrotinib; neratinib; Imatinib Mesylate; palbociclib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Standard treatment Group (No Intervention): Patients with rare tumours in this group will undergo standard treatment in accordance with the leading domestic and international guidelines (NCCN/ESMO/CSCO/CACA) and clinical trial.
- Criteria-Fulfilled ICF Group (Experimental): Intervention in this group is to perform PDOs culture and drug screening of lesions from patients with rare tumours who failed to standard treatment and fully meet the inclusion and exclusion criteria. The MTB will review the results of the drug screening and NGS, and subsequently determine the personalised chemotherapy, targeted or immunological agents.
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Epirubicin; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Cisplatin; Drug: Irinotecan; Drug: Fluorouracil; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Durvalumab; Drug: Atezolizumab; Drug: Sintilimab; Drug: Tislelizumab; Drug: Camrelizumab; Drug: Toripalimab; Drug: Serplulimab; Drug: Adebrelimab; Drug: Envafolimab; Drug: Osimertinib; Drug: Alectinib; Drug: Vemurafenib; Drug: Pamiparib; Drug: Pyrotinib; Drug: Imatinib; Drug: Palbociclib; Drug: Savolitinib; Drug: Entrectinib
- Compassionate-Use ICF Group (Experimental): Patients with rare tumours who failed to standard treatment and do not meet the requisite criteria (e.g. active hepatitis B, underlying disease in the exclusion criteria, symptomatic brain metastases) will provide informed consent and undergo PDOs culture and drug screening. The MTB will review the results of the drug screening and NGS, and subsequently determine the personalised chemotherapy, targeted or immunological agents.
  Interventions: Drug: Albumin-Bound Paclitaxel; Drug: Epirubicin; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Cisplatin; Drug: Irinotecan; Drug: Fluorouracil; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Durvalumab; Drug: Atezolizumab; Drug: Sintilimab; Drug: Tislelizumab; Drug: Camrelizumab; Drug: Toripalimab; Drug: Serplulimab; Drug: Adebrelimab; Drug: Envafolimab; Drug: Osimertinib; Drug: Alectinib; Drug: Vemurafenib; Drug: Pamiparib; Drug: Pyrotinib; Drug: Imatinib; Drug: Palbociclib; Drug: Savolitinib; Drug: Entrectinib
- RWS ICF Group (Experimental): Patients with rare tumours who failed to standard treatment will be included in a real-world study cohort and receive clinically conventional treatment if they do not undergo PDOs culture and NGS testing successfully or are unwilling to base their treatment on the results of PDOs and NGS for various reasons.
  Interventions: Drug: Other

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel — Albumin-Bound Paclitaxel 260mg/m2,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with albumin-bound paclitaxel if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Abraxane
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Epirubicin — Epirubicin 90mg/m2,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with epirubicin if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Ellence
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Gemcitabine — Gemcitabine 1000mg/m2,D1,D8,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with gemcitabine if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Gemzar
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Vinorelbine — Vinorelbine 25-30mg/m2,D1,D8,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with vinorelbine if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Navelbine; Vumon
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Cisplatin — Cisplatin 90mg/m2,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with cisplatin if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Platinol
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Irinotecan — Irinotecan 125mg/m2,D1,D8,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with irinotecan if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Camptosar
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Fluorouracil — Fluorouracil 600mg/m2,D1-5,q3w Patients with advanced rare tumours who failed to standard treatment will be administrated with fluorouracil if PDOs show the highest response to this drug under the guidance of MTB.
  Other Names: Adrucil; 5-FU
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Nivolumab — Nivolumab 3mg/kg,q2w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with nivolumab under the guidance of MTB.
  Other Names: Opdivo
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Pembrolizumab — Pembrolizumab 200mg,q2w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with pembrolizumab under the guidance of MTB.
  Other Names: Keytruda
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Durvalumab — Durvalumab 10mg/kg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with durvalumab under the guidance of MTB.
  Other Names: Imfinzi
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Atezolizumab — Atezolizumab 1200mg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with atezolizumab under the guidance of MTB.
  Other Names: Tecentriq
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Sintilimab — Sintilimab 200mg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with sintilimab under the guidance of MTB.
  Other Names: Tyvyt
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Tislelizumab — Tislelizumab 200mg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with tislelizumab under the guidance of MTB.
  Other Names: Baizean
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Camrelizumab — Camrelizumab 200mg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with camrelizumab under the guidance of MTB.
  Other Names: AiRuiKa
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Toripalimab — Toripalimab 240kg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with toripalimab under the guidance of MTB.
  Other Names: Tuoyi
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Serplulimab — Serplulimab 3mg/kg,q2w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with serplulimab under the guidance of MTB.
  Other Names: Hansizhuang
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Adebrelimab — Adebrelimab 20mg/kg,q3w Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with adebrelimab under the guidance of MTB.
  Other Names: Abesive
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Envafolimab — Envafolimab 150mg,qw Patients with advanced rare tumours who failed to standard treatment carrying no targeted alterations will be administrated with envafolimab under the guidance of MTB.
  Other Names: Epkinly
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Osimertinib — Osimertinib 80mg,qd Patients with advanced rare tumours who failed to standard treatment carrying EGFR mutations will be administrated with osimertinib under the guidance of MTB.
  Other Names: Tagrisso
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Alectinib — Alectinib 600mg,bid Patients with advanced rare tumours who failed to standard treatment carrying ALK fusion will be administrated with alectinib under the guidance of MTB.
  Other Names: Alecensa
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Vemurafenib — Vemurafenib 960mg,bid Patients with advanced rare tumours who failed to standard treatment carrying BRAF V600E mutation will be administrated with vemurafenib under the guidance of MTB.
  Other Names: Zelboraf
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Pamiparib — Pamiparib 60mg,bid Patients with advanced rare tumours who failed to standard treatment carrying BRCA1/2 mutation will be administrated with pamiparib under the guidance of MTB.
  Other Names: Balversa
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Pyrotinib — Pyrotinib 400mg, qd Patients with advanced rare tumours who failed to standard treatment carrying HER-2 mutation or HER-2 over expression/amplification will be administrated with Pyrotinib under the guidance of MTB.
  Other Names: Nerlynx
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Imatinib — Imatinib 400mg, qd Patients with advanced rare tumours who failed to standard treatment carrying CKIT mutation will be administrated with imatinib under the guidance of MTB.
  Other Names: Gleevec
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Palbociclib — Palbociclib 125mg, 21/7 dosing schedule Patients with advanced rare tumours who failed to standard treatment following HR(+)/HER-2(-) will be administrated with palbociclib under the guidance of MTB.
  Other Names: Ibrance
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Savolitinib — Savolitinib 300mg, qd Patients with advanced rare tumours who failed to standard treatment carrying C-MET mutation will be administrated with savolitinib under the guidance of MTB.
  Other Names: Orpathys
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Entrectinib — Entrectinib 600mg, qd Patients with advanced rare tumours who failed to standard treatment carrying ROS-1 fusion or NTRK fusion will be administrated with entrectinib under the guidance of MTB.
  Other Names: Rozlytrek
  Arms: Compassionate-Use ICF Group; Criteria-Fulfilled ICF Group
Drug: Other — Patients with advanced rare tumours who failed to standard treatment in RWS ICF Group will be administrated with empirical chemotherapy(e.g., "Albumin-Bound Paclitaxel", "Epirubicin", "Gemcitabine", "Vinorelbine", "Cisplatin", "Irinotecan", "Fluorouracil"), immunological(e.g., "Nivolumab", "Pembrolizumab", "Durvalumab", "Atezolizumab", "Sintilimab", "Tislelizumab", "Camrelizumab", "Toripalimab", "Serplulimab","Adebrelimab","Envafolimab") or targeted drugsl(e.g., "Osimertinib", "Alectinib", "Vemurafenib", "Vemurafenib", "Pyrotinib", "Imatinib", "Palbociclib", "Savolitinib", "Entrectinib")treatments.
  Arms: RWS ICF Group

SUMMARY:
The objective of this Phase II, open-label, multicenter, non-randomised controlled clinical trial is to guide precision treatment for patients with rare tumours based on Patient-Derived Organoids/Next-Generation Sequencing drug screening.

DETAILED DESCRIPTION:
Rare tumours, defined as those with an annual incidence rate of less than 2.5/100,000 according to the data from the National Cancer Registry of the National Cancer Center of China, represent a significant unmet medical need due to the lack of high-level evidence-based clinical practice guidelines and standard regimens. Patient-Derived Organoids(PDOs), which preserves the histologic and genetic characteristics of patients; tumours, have demonstrated predictive value of clinical outcomes. Prior studies have shown that PDOs-based drug screens can predict treatment response with high sensitivity and specificity.The investigators thus propose the study: A Phase II Clinical Study on Precision Treatment of Rare Tumours in China Guided by Patient-Derived Organoids and Next-Generation Sequencing. Investigators aim to determine clinical efficacy of PDOs/NGS-guided precision treatment in patients with rare tumours. After tumour samples were collected, drug screening using PDOs and NGS will be conducted. Molecular Tumor board(MTB) will review the results and develop an individualised treatment regimens. Primary endpoint of this study is objective response rate (ORR). Secondary endpoints include disease control rate (DCR), progression-free survival (PFS), overall survival (OS) and duration of response (DoR).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, the age at the time of signing the informed consent is no less than 18 years old;
2. Patients with advanced or metastatic rare solid tumor confirmed by histological confirmed;
3. ECOG score is 0 or 1;
4. Expected survival ≥12 weeks;
5. According to Response Evaluation Criteria in Solid Tumor (RECIST 1.1), there is at least one imaging measurable lesions, which has not previously undergone radiotherapy or with obvious disease progress after radiotherapy;
6. Surgical specimens of paired tumor tissue and adjacent normal tissue, or fresh biopsy tissue samples or ≥500ml serous cavity effusion with positive pathological cytological examination must be provided. These specimens must be obtained without prior exposure to any other anti-tumor treatment, systemic anti-infection treatment, vaccination, et al. and are intended for organoid culture;
7. Must have a primary or metastatic paraffin-embedded tissue (without radiotherapy) other than bone metastatic lesions before enrollment (within 2 years, 15-20 sheets, 4-6μm thick white slices, of which 5 need to be glued and baked ) and peripheral blood samples for NGS gene testing. If NGS results are already available but sufficient paraffin-embedded tissue cannot be provided, investigator are allowed the decision to enroll subjects according to the specific situation;
8. In the condition that the primary lesions biopsy specimen has been provided, if the metastatic lesion is able to be biopsied(determined by investigator), it is suggested to keep the specimen for pathological testing and provide fresh tissue specimen;
9. After the progression of the subject's disease, if conditions permit(determined by investigator), fresh tissue samples shall be obtained from the same biopsy lesions and the metastasis lesions of the previously obtained samples;
10. Toxic and side effects caused by previous treatment need to be restored to ≤ Grade 1 or returned to the baseline value (NCI-CTCAE version 5.0, except for hair loss);
11. Negative pregnancy test (only applicable for women with childbearing potential). No childbearing potential is defined as being postmenopausal for longer than one year or having undergone surgical sterilization or hysterectomy;
12. All patients (male and female) agree to use an effective form of contraceptive measures during the treatment and within 8 weeks after the end of treatment;
13. Signed, written informed consent of volunteers that join the group shall follow the trial treatment plan, follow-up plan and cooperate to observe the adverse events and efficacy.

Exclusion Criteria:

1. No patient lesions available for organoid model construction;
2. History of interstitial lung disease or radiation pneumonitis of any type;
3. Central Nervous System (CNS) metastases with brain metastases-related symptoms, which is not stable in neurology, or need to increase steroid dosage to control CNS disease. (Note: Patients with controlled CNS metastasis are eligible to participate in this study);
4. Current uncontrollable third cavity effusion, such as a large amount of pleural effusion，ascites , or pericardial effusion;
5. Major surgical operations or incomplete healing of injury within 4 weeks prior to study treatment's first administration and chest radiotherapy of > 30 Gy within 6 months;
6. History of receiving other investigational drugs within 14 days or 5 half-lives (whichever is longer) prior to the first administration;
7. History of receiving live vaccine within 30 days prior to the first administration. Seasonal influenza vaccines that do not contain live viruses are allowed;
8. Current active infection requiring systemic treatment (antibiotics); or any of the following:

   1. HIV positive or known history of acquired immunodeficiency syndrome;
   2. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection is defined as HBsAg positive and the number of HBV DNA copies exceeds the upper limit of normal value, or HCV AB positive;
   3. Active tuberculosis (with exposure history or positive tuberculosis test; with clinical and / or imaging manifestations);
   4. Positive antibody of Treponema Pallidum
9. Current evidenced uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [still greater than or equal to CTCAE Grade 3 hypertension after drug treatment]);
10. History of myocardial infarction, coronary artery / peripheral artery bypass or cerebrovascular accident within 3 months;
11. Diagnosed with a second type of malignant tumor within 5 years before the first diagnosis of a rare solid tumor (excluding completely resected basal cell carcinoma, bladder carcinoma in situ, cervical carcinoma in situ);
12. History of receiving of any organ transplantation, including allogeneic stem cell transplantation. Transplantation without immunosuppression (corneal transplantation, hair transplantation) is excluded;
13. Cardiovascular disease or symptom includes any of the following:

    1. History of Congestive Heart Failure requiring treatment and of New York Heart Association class III / IV CHF (see Appendix 3) ;
    2. Current ventricular arrhythmia requiring antiarrhythmic drugs treatment, or uncontrollable or unstable arrhythmia;
    3. Severe conduction disorder (such as grade II or III AV block);
    4. Angina requiring treatment;
    5. QT interval (QTC) of 12 lead ECG is ≥ 450 ms in male and ≥ 470 MS in female;
    6. History of congenital long QT syndrome, congenital short QT syndrome, torsade de pointe or pre-excitation syndrome;
    7. History of LVEF decline to below 50% determined by echocardiography or MUGA scan;
    8. History of myocardial infarction in the past 6 months.
14. Inadequate bone marrow reserve or organ function;
15. Pregnant or lactating women;
16. History of swallowing dysfunction, active gastrointestinal disease or other diseases that significantly affect the absorption, distribution, metabolism and excretion of oral drugs. The patients with history of subtotal gastrectomy. (Note: this standard is not applicable to the sub schemes with the investigational drug as injection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment to the end of treatment at 8 weeks
  The percentage of patients with a confirmed investigator-assessed complete or partial response according to Response Evaluation Criteria In Solid Tumours (RECIST) 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From enrollment to the end of treatment at 8 weeks
  The percentage of evaluable patients who achieve confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (lasting for ≥ 8 weeks).
Progression free survival (PFS) | From enrollment to the end of treatment at 8 weeks
  Time from the first dose of treatment until the first documentation of disease progression (PD) or death from any cause, whichever occurs first.
Overall survival (OS) | From enrollment to the end of treatment at 8 weeks
  Time from the first dose of treatment until the death of the patient from any cause.
Duration of response (DOR) | From enrollment to the end of treatment at 8 weeks
  Time from the first tumor assessment showing a Complete Response (CR) or Partial Response (PR) to the first occurrence of disease progression (PD) or death before PD in subjects who achieved CR or PR, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: shunbin wang, Doctor, Study Chair — Peking University Shenzhen Hospital

IPD SHARING:
Plan to Share IPD: Undecided